CLINICAL TRIAL: NCT06751056
Title: Neck Traction to Reduce Gabaergic Medication Use for Neuropathic Itch- A Pilot Study
Brief Title: Cervical Traction to Reduce Gabaergic Medication Use for Neuropathic Itch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David L. Swanson, Professor of Dermatology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-003108
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cervical Traction Group (Experimental): Patients who are on a stable dosage of gabapentin or pregabalin for scalp, arm or upper back pruritus without primary rash
  Interventions: Device: Cervical Traction Device

INTERVENTIONS:
Device: Cervical Traction Device — Participants will use their home neck traction devices daily for 12 weeks, while continuing their prescriptions for gabapentin or pregabalin.
  At study initiation and every 2 weeks thereafter for a total of 12 weeks, they will receive an electronic survey assessing their itch score. Based on survey results, they will receive a call from the study team to adjust their dosage of gabapentin or pregabalin by up to 33%.

SUMMARY:
The purpose of this study is to determine if cervical traction is an effective treatment to reduce GABAergic medication use for scalp, arm, and upper back neuropathic itch.

ELIGIBILITY:
Inclusion Criteria

* Persons with scalp, arm, and upper back pruritus without primary skin lesions.
* Persons 18 or older.
* Person on a stable dosage of gabapentin or pregabalin over the preceding 4 week period.
* Persons willing and able to comply with clinic visits and study-related procedures.
* Persons willing and able to understand and complete study-related questionnaires.
* Persons willing and able to provide voluntary signed informed consent.

Exclusion Criteria

* Primary skin lesions driving scalp, arm, or upper back pruritus.
* A history of spinal surgery or other conditions (acute or traumatic spinal injury, spinal instability, spinal fracture, rheumatoid arthritis, metastatic disease to the spine, spinal cord compression, active infections of the head and neck) that would make neck traction contraindicated.
* Unable to comfortably lay down on the floor and get back up without assistance.
* Medical conditions in which gabapentin and/or pregabalin is contraindicated.
* Current enrollment in physical therapy with exercises addressing the cervical spine.
* Planned or anticipated use of any prohibited medications or procedures during study treatment.
* Presence of skin comorbidities that may interfere with study assessments.
* Currently pregnant or breastfeeding or plans to become pregnant or breastfeed during the participation in the study. Persons of childbearing age who are not on reliable contraception will be considered on a case-by-case basis.

  o Participants of childbearing age who are not on reliable contraception (hormonal contraceptive pills, patch, or ring, intrauterine device, subdermal hormonal implant, tubal ligation, depot medroxyprogesterone injections) will be required to complete monthly urine pregnancy tests.
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study. Examples include, but are not limited to, a short life expectancy, persons with uncontrolled diabetes (HbA1c ≥ 9%), cardiovascular conditions (e.g. stage III or IV cardiac failure), severe renal conditions (e.g. patients on dialysis), debilitating neurological conditions (e.g. demyelinating diseases), active major autoimmune diseases (e.g. lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), or other severe endocrinological, gastrointestinal, hepatobiliary, metabolic, pulmonary, or lymphatic diseases. The specific justification for persons excluded under this criterion will be noted in study documents.
* Any other medical or psychological condition (including relevant laboratory abnormalities at screening) that, in the opinion of the investigator, may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study patient as a result of his/her participation in this clinical trial, may make participation unreliable, or may interfere with study assessments. The specific justification for persons excluded under this criterion will be noted in study documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in GABAergic medication usage | Baseline, 12 weeks
  Reported as percentage of reduction in dosage of gabapentin or pregabalin after 12 weeks of home neck traction.

SECONDARY OUTCOMES:
Pruritus Severity Score | Baseline, 14 days, 28 days, 42 days, 56 days, and 72 days
  A 12-item questionnaire assessing different aspects of pruritus. The items are grouped into five domains: pruritus intensity, pruritus extent, frequency and duration of pruritus, impact of pruritus on daily activities and mood, and assessment of scratching. Total scoring ranges from 3 (the lowest pruritus intensity) to 22 points (the highest pruritus intensity).

CONTACTS AND LOCATIONS:
Overall Officials: David Swanson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials